CLINICAL TRIAL: NCT04632784
Title: Prospective Multicentre Clinical Trial With the Artiflex Presbyopic (Artiplus), an Iris-fixated Multifocal Intraocular Lens for the Correction of Presbyopia in Phakic Eyes
Brief Title: Clinical Trial With Artiflex Presbyopic (Artiplus)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ophtec BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP01000816
Record Dates: First submitted 2020-10-30; First posted 2020-11-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Presbyopia; Ametropia; Refractive Errors; Myopia; Hyperopia
Keywords: Artiflex Presbyopic; iris-fixated; phakic intraocular lens; PIOL; Ophtec; Artiplus
MeSH Terms: conditions — Presbyopia; Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artiflex Presbyopic (Artiplus) (Experimental): 49 subjects have received the Artiflex Presbyopic lens (Artiplus) bilaterally and will be followed for 3 years.
  Interventions: Device: Artiflex Presbyopic (Artiplus) implantation

INTERVENTIONS:
Device: Artiflex Presbyopic (Artiplus) implantation — Implantation of iris-fixated multifocal Artiflex Presbyopic IOL (Artiplus)

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and safety of the multifocal Artiflex Presbyopic (Artiplus) intraocular lens.

DETAILED DESCRIPTION:
The study is a prospective, open-label, single-arm, and multicentre clinical investigation with three years of follow-up. Artiflex Presbyopic (Artiplus) is a phakic intraocular lens to be implanted in the anterior chamber, intended for adult subjects and indicated for the optical correction of presbyopia and spherical error requiring a correction.

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic adult
* Potential for binocular vision
* Subject wishes to be spectacle independent for near and far vision
* Refractive error that can be corrected with correction at PIOL plane from +2.0 to -15.0 D
* Subject requiring a presbyopic correction Patients with reading glasses of minimum +1D.
* Stable refraction (±0.75 D), as expressed by manifest refraction spherical equivalent (MRSE) for a minimum of 12 months prior to surgery, verified by consecutive refractions and/or medical records or prescription history
* Expected best corrected visual acuity of 0.2 logMAR (0.63 Snellen decimal) or better after lens implantation
* Current contact lens wearer should demonstrate a stable refraction (± 0.5 D), expressed as subjective refraction spherical equivalent, on two consecutive examination dates performed at least 7 days apart. Before the first refraction, the contact lens wearer should not have worn lenses for at least 2 weeks in case of rigid and toric contact lenses, or 3 days for spherical soft contact lenses.
* Any subject, who is expected to have a residual postoperative cylindrical refractive error of below 0.75 D
* Ability to give informed consent
* Availability, willingness and sufficient cognitive awareness and physical ability to comply with examination procedures throughout the entire duration of the study

Exclusion Criteria:

Pre-existing pathology or physiology which may be aggravated by the implant or where the implant may interfere with the possibility of examining or treating disease:

* Preoperative ocular or systemic condition or medication use that would be expected to present undue risk to the subject, that can predispose for future complications or confound the outcome(s) of the study. E.g. the systemic use of alpha-1a adrenergic receptor antagonists was suggested to increase the occurrence of intraoperative floppy iris syndrome, alter iris morphology - or more specifically reduce iris thickness at the site of potential IOL enclavation - and increase postoperative endothelial cell loss.
* Previous ocular surgery which might affect the outcome of the study
* Concurrent participation or participation during the last 30 days in another drug or device investigation
* Secondary surgical procedure planned during the first 6 months of the study (e.g. laser treatment to correct astigmatism)
* Amblyopia
* Preoperative anterior chamber depth measurement of below 3.0 mm for subjects < 40 years old and 2.8 mm for subjects > 40 years old. Anterior chamber depth is being measured from corneal endothelium to the anterior pole of the crystalline lens. This will result in a critical distance between PIOL and endothelium of 1.5 mm or more as simulated with anterior segment imaging.
* White-to-white smaller than 10.5 mm
* Subjects not meeting the age specific minimum preoperative endothelial cell density as defined below:

  31 to 35 years of age 2400 cells/mm2; 36 to 45 years of age 2200 cells/mm2; > 45 years of age 2000 cells/mm2
* Corneas with high rates of polymegethism (a coefficient of variation over 0.40) and pleomorphism (the presence of less than 50% hexagonal cells).
* Abnormal iris (e.g. convex, bulging or volcano shaped iris)
* Crystalline lens rise of 600 µm or more
* Abnormal cornea (keratoconus, opaque cornea, corneal scars, post corneal transplant, corneal dystrophy, or other)
* Ocular surface conditions which might influence the quality of vision and affect the outcome of the study
* Abnormal pupil (e.g. nonreactive, fixed)
* Ectopic pupil
* Pupil in photopic light conditions smaller than 2.6 mm
* Pupil in scotopic light conditions greater than 7.0 mm
* High preoperative intraocular pressure (>21 mm Hg)
* Cataract of any grade
* Glaucoma or family history of glaucoma (dependent on the evaluation of physician)
* Diabetes or diabetic retinopathy
* Acute or chronic inflammation
* Chronic or recurrent uveitis or family history of the same condition
* Retinal detachments or family history of retinal detachments
* Corticosteroid responder
* Pregnant or nursing
* Unstable refraction (≥ 0.5D of variability in refraction over the last 12 months)
* Aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Improvement in monocular and binocular uncorrected near visual acuity (UNVA) | 3 years
  * Percentage of eyes that achieve UNVA of 0.3 logMAR or better
  * Percentage of eyes that achieve UNVA of 0.0 logMAR or better
Improvement in monocular and binocular corrected near visual acuity (CNVA) | 3 years
  * Percentage of eyes that achieve CNVA of 0.3 logMAR or better
  * Percentage of eyes that achieve CNVA of 0.0 logMAR or better
Improvement in monocular and binocular distance corrected near visual acuity (DCNVA) | 3 years
  * Percentage of eyes that achieve DCNVA of 0.3 logMAR or better
  * Percentage of eyes that achieve DCNVA of 0.0 logMAR or better
Improvement in monocular and binocular uncorrected intermediate visual acuity (UIVA) | 3 years
  * Percentage of eyes that achieve UIVA of 0.3 logMAR or better
  * Percentage of eyes that achieve UIVA of 0.0 logMAR or better
Improvement in monocular and binocular distance corrected intermediate visual acuity (DCIVA) | 3 years
  * Percentage of eyes that achieve DCIVA of 0.3 logMAR or better
  * Percentage of eyes that achieve DCIVA of 0.0 logMAR or better
Improvement in monocular and binocular uncorrected distance visual acuity (UDVA) | 3 years
  Percentage of eyes that achieve UDVA of 0.3 logMAR or better Percentage of eyes that achieve UDVA of 0.0 logMAR or better
Improvement in monocular and binocular corrected distance visual acuity (CDVA) | 3 years
  * Percentage of eyes that achieve CDVA of 0.3 logMAR or better
  * Percentage of eyes that achieve CDVA of 0.0 logMAR or better
Defocus evaluation | 3 years
  Binocular defocus evaluation will be obtained by using the best-corrected distance refraction and then defocusing the image in 0.5 D increments from +1.5 to -5.0 D
Predictability of the manifest refraction spherical equivalent (MRSE) | 3 years
  The absolute difference between the actually obtained MRSE and the target MRSE
Predictability of the manifest refraction spherical equivalent (MRSE) | 3 years
  The percentage of eyes that achieves a MRSE of less than or equal to 0.5 D difference between the actual and target MRSE
Predictability of the manifest refraction spherical equivalent (MRSE) | 3 years
  The percentage of eyes that achieves a MRSE of less than or equal to 1.0 D difference between the actual and target MRSE
Stability of manifest refraction spherical equivalent (MRSE) | 3 years
  Mean change in MRSE between visits as determined by a paired analysis
Stability of manifest refraction spherical equivalent (MRSE) | 3 years
  The percentage of eyes that achieves a change in MRSE of less than or equal to 0.5 D between two consecutive refraction measurements
Stability of manifest refraction spherical equivalent (MRSE) | 3 years
  The percentage of eyes that achieves a change in MRSE of less than or equal to 1.0 D between two consecutive refraction measurements
Evaluation of visual disturbances using a validated questionnaire | 3 years
  Assessing the percentage of subjects who experience different visual disturbances, by means of questionnaire
Evaluation of visual disturbances using a validated questionnaire | 3 years
  Assessing the occurrence of the different visual disturbances by means of questionnaire
Evaluation of visual disturbances using a validated questionnaire | 3 years
  Assessing the severity of the different visual disturbances by means of questionnaire
Evaluation of visual disturbances using a validated questionnaire | 3 years
  Assessing the bothersomeness of the different visual disturbances by means of questionnaire
Evaluation of visual disturbances using a validated questionnaire | 3 years
  Assessing the time of onset of visual disturbances by means of questionnaire
Satisfaction questionnaire | 3 years
  * Percentage of subjects that is satisfied with the overall procedure
  * Percentage of subjects that is satisfied with uncorrected near vision
  * Percentage of subjects that is satisfied with uncorrected intermediate vision
  * Percentage of subjects that is satisfied with uncorrected distance vision
Endothelial cell density | 3 years
  Comparison of the preoperative and postoperative endothelial cell density
Endothelial cell density | 3 years
  Endothelial cell loss over time
Endothelial cell density | 3 years
  Additionally, a comparison between the scientific literature reported naturally occurring endothelial cell loss over time (approx. 0.6% per year; Bourne et al., 1997) and the study observed cell loss will be performed
Adverse event (AEs) / complication rates | 3 years
  * Cumulative numbers of adverse events, e.g. cystoid macular edema (CME), hypopyon, endophthalmitis, lens dislocation, pupillary block, retinal detachment, necessary secondary surgical interventions
  * Cumulative numbers of adverse events persistently present, e.g. corneal stroma edema, cystoid macular edema, iritis, raised intraocular pressure (IOP) requiring treatment, lens deposits
  * The occurrence of adverse events will be compared to and should not exceed the reference safety and performance endpoint (SPE) rates as defined by ISO 11979-7:2018, Annex E, table E.1

CONTACTS AND LOCATIONS:
Overall Officials: J. Guell, MD, Principal Investigator — Instituto de Microcirugía Ocular, Barcelona, Spain
Locations (7):
- South Korea (3):
  - GM st. Mary's Eye clinic, Busan
  - Nune Eye Hospital Daegu, Seoul
  - SU Yonsei Eye Clinic, Seoul
- Spain (4):
  - ICQO, Bilbao, Biscay
  - IMO, Barcelona, Catalonia
  - Hospital San Rafael, Madrid
  - CIMO, Seville